CLINICAL TRIAL: NCT07178184
Title: Evaluating the Efficacy and Safety of Modified Qing-Zao-Jiu-Fei Decoction on Pneumoconiosis Patients: A Randomized, Double-blinded, Placebo-Controlled Trial
Brief Title: Evaluating the Efficacy and Safety of Modified Qing-Zao-Jiu-Fei Decoction on Pneumoconiosis Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, XIAN Yanfang, Prof. XIAN Yanfang, Assistant professor, School of Chinese Medicine, Faculty of Medicine, The Chinese University of Hong Kong, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCFB study
Record Dates: First submitted 2025-09-09; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Pneumoconiosis
Keywords: RCT; Chinese Medicine; Pneumoconiosis
MeSH Terms: conditions — Pneumoconiosis

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, double-blind, placebo-controlled study to investigate the beneficial efficacy and safety of Modified Qing Zao Jiu Fei Decoction (MQZJFD) on pneumoconiosis patients will be carried out in two Integrative Medical Centres (Shatin and Wan Chai), CUHK (IMCs-SCM), the CUHK-Chinese Medicine Specialist Clinic cum Teaching and Research Centre (CUHK-CMSCTRC) at the School of Chinese Medicine, CUHK, and the Centre for Clinical Trials on Chinese Medicine (CCTCM), Institute of Chinese Medicine, CUHK. Participants will be randomized into one of the two groups (MQZJFD treatment group or placebo control group), and both undergo a consultation process by the Chinese Medicine practitioner (CMP). Eligible participants will be randomized and receive either MQZJFD granules or placebo granules for 16 weeks followed by post-treatment visits at week 20. The study will last for 20 weeks with a treatment period of 16 weeks plus a follow-up period of 4 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Qing-Zao-Jiu-Fei Decoction (MQZJFD) (Experimental): A chinese medicine formular
  Interventions: Drug: Modified Qing-Zao-Jiu-Fei Decoction (MQZJFD)
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modified Qing-Zao-Jiu-Fei Decoction (MQZJFD) — MQZJFD is the core formula in this clinical study and consists of the 11 following herbs: Mori Folium 9g, Plaster stone 9g, Trichosanthis Fructus 9g, Ophiopogyonis Radix 6g, Armeniacae Semen Amarum 6g, Fritillariae Thunbergii Bulbus 6g, Eriobotryae Folium 6g, Ginseng Radix et Rhizoma 3g, Semen Sesami Nigrum 3g, Asini Corii Colla 3g, Glycyrrhizae Radix et Rhizoma 3g.
  The formula will be prepared with single concentrated herbal granules (1 g of single concentrated herbal granule equates to 5 g of original dry herbs, except for Ophiopogyonis Radix whose ratio will be that 1 g of single concentrated herbal granule equals to 3 g of original dry herb, and Asini Corii Colla whose ratio will be that 1 g of single concentrated herbal granule equals to 1 g of original dry herb). The herbal granules will be provided by a Good Manufacturing Practice (GMP)-accredited supplier.
  Arms: Modified Qing-Zao-Jiu-Fei Decoction (MQZJFD)
Drug: Placebo — The placebo granules consists of an inert substance made of starch filler, silica coating, flavor and coloring. Its appearance is unidentifiable to the real intervention drug. The placebo granules is also manufactured under GMP standards. To ensure blinding, the MQZJFD granules and placebo granules will be indistinguishable in appearance, smell and flavor.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to investigate the beneficial efficacy and safety of Chinese medicine formula Modified Qing Zao Jiu Fei Decoction (MQZJFD) on pneumoconiosis patients. Participants will be randomized into one of the two groups (MQZJFD treatment group or placebo control group), and both undergo a consultation process by the Chinese Medicine practitioner (CMP). Eligible participants will be randomized and receive either MQZJFD granules or placebo granules for 16 weeks followed by post-treatment visits at week 20. The study will last for 20 weeks with a treatment period of 16 weeks plus a follow-up period of 4 weeks.

ELIGIBILITY:
Inclusion criteria

1. Aged 20-85;
2. Patients with pneumoconiosis (Confirmed case of pneumoconiosis by Pneumoconiosis compensation fund board);
3. Agree to undergo blood test and willing to complete questionnaires and take medication as scheduled; and
4. Willing to provide written informed consent.

Exclusion criteria

1. Patient with the following Chinese medicine syndromes/patterns according to Chinese medicine theory: dampness, lung deficiency and coldness, or Yang deficiency according to Chinese medicine theory;
2. Patients receiving Chinese medicine in a regular pattern within the past 2 weeks;
3. Patients with chronic co-morbidities such as other fibrotic lung diseases in addition to pneumoconiosis and/or co-existing heart disease;
4. Patients with a medical history of malignancy within the past 5 years;
5. Patients with a medical history of any serious diseases such as severe kidney and liver impairments, autoimmune disease, thyroid disease, Hodgkin's disease, lymphoma and leukemia;
6. Patients with known severe cognitive and mental disorders;
7. Documented pregnancy or lactation; or
8. Patients allergic to the drug used in this study.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of 6-minute Walk Test (6MWT) at weeks 4, 8, 12, 16 and 20. | Baseline, weeks 4, 8, 12, 16 and 20.
  The 6MWT, developed by Balke in 1963, is one of the tests widely used to assess functional exercise capacity evaluated by measuring the distance walked during 6 min. The test is easy to administer and is better tolerated and more reflective of the activities of daily living than other walk tests. Most activities of daily life usually are performed at a submaximal level of exertion, so the 6MWT seems to better reflect the functional exercise level for daily physical activities. Accordingly, the 6MWT would be a good estimation tool for objective health and assessment in pneumoconiosis and the test will be carried out according to the standards of the American Thoracic Society . The 6MWT will be conducted by trained investigators or research assistants.

SECONDARY OUTCOMES:
Change of St. George's Respiratory Questionnaire - Hong Kong version (SGRQ-HK) at weeks 4, 8, 12, 16 and 20 | Baseline, weeks 4, 8, 12, 16 and 20
  SGRQ is a disease-specific instrument designed for, and commonly applied in, patients with chronic obstructive lung disease (COPD). The SGRQ has three components: (1) Symptom, measuring respiratory symptoms; (2) Activity, measuring impairment of mobility or physical activity, and (3) Impact, measuring the psychosocial impact of disease. It has a Chinese version validated in Hong Kong (the SGRQ-HK), which has been applied in two Hong Kong studies of pneumoconiosis.
Change of Pittsburgh Sleep Quality Index (PSQI) at weeks 4, 8, 12, 16 and 20 | Baseline, weeks 4, 8, 12, 16 and 20
  PSQI measures the quality and pattern of sleep in older adult by measuring seven domains in 19 questions: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication and daytime dysfunction over the last month. The scoring is 0-3 on a Likert scale.
Change of Hospital anxiety and depression scale (HADS) at weeks 4, 8, 12, 16 and 20 | Baseline, weeks 4, 8, 12, 16 and 20
  The HADS, developed by Zigmond and Snaith in 1983, is a 14-item self assessment questionnaire commonly used to measure the severity of anxiety and depression in individuals undergoing medical care. It is now widely used in clinical and research settings. Many studies conducted around the world have confirmed its validity in community and primary care medical practice. HADS is often used to evaluate the mental health of patients with physical or chronic illnesses. The HADS questionnaire has 7 questions for anxiety and 7 questions for depression, with a scale of 0-3. Higher scores indicate higher levels of anxiety or depression.
Change of COPD Assessment Test (CAT) at weeks 4, 8, 12, 16 and 20 | Baseline, weeks 4, 8, 12, 16 and 20
  The CAT is a tool used to assess the severity of symptoms in patients with COPD, it can also be used in patients with pneumoconiosis. It consists of eight questions to assess the severity of symptoms and effects of COPD in daily life. These questions relate to dyspnoea, cough, sputum retention, chest pain, sleep quality, energy levels, mobility and anxiety. Each problem is rated on a scale of 0 to 5, the higher the score the more severe the symptoms.
Change of Patient Global Impression of Change (PGIC) at weeks 4, 8, 12, 16, 20 | Baseline, weeks 4, 8, 12, 16, 20
  Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", or "very much worse".
Frequency of patients suffering from colds after baseline | From baseline to week 20
Incidence of patient hospitalization during the trial | From baseline to week 20
Change of the measurement of the body weight of patients | From baseline to week 20
Adverse events related to study treatment | From baseline to week 20

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://clinicaltrials.gov